CLINICAL TRIAL: NCT07393165
Title: The Effect of Levothyroxine Treatment on Cardiac Function in Children With Subclinical Hypothyroidism
Brief Title: Levothyroxine Treatment on Cardiac Function in Children With Subclinical Hypothyroidism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Zeinab Ebraheem Amin Elshareef, Resident of Pediatrics, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36264MS959/5/25
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Levothyroxine; Cardiac Function; Children; Subclinical Hypothyroidism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Children with subclinical hypothyroidism who will receive L-thyroxine treatment in a dose of 2μg/kg/d (the smallest dose can be given) and the dose will be titrated every 4 weeks until a normal thyroid-stimulating hormone (TSH) level is maintained.
  Interventions: Drug: L-thyroxine
- No treatment group (No Intervention): Children with subclinical hypothyroidism who will receive no treatment.

INTERVENTIONS:
Drug: L-thyroxine — Children with subclinical hypothyroidism who will receive L-thyroxine treatment in a dose of 2μg/kg/d (the smallest dose can be given) and the dose will be titrated every 4 weeks until a normal thyroid-stimulating hormone (TSH) level is maintained.
  Arms: Treatment group

SUMMARY:
This study aims to evaluate the effect of the treatment with levothyroxine on cardiac function in children with subclinical hypothyroidism.

DETAILED DESCRIPTION:
Subclinical hypothyroidism (SH) is a branch of hypothyroidism which is characterized by increased thyroid stimulating hormone (TSH) and normal thyroxine (T4).

Inadequate serum thyroid hormone levels impair cardiac function and may result in multiple cardiovascular risk factors, such as endothelial dysfunction, increased intima-media thickness, increased vascular resistance, and pericardial effusion.

ELIGIBILITY:
Inclusion Criteria:

* Age from 4 to 15 years.
* Both sexes.
* Patients with stable elevated thyroid-stimulating hormone (TSH) ≥ 4.5 mIU/L with normal free T4 and ft3 in different measurement 4 - 6 weeks apart.

Exclusion Criteria:

* Overweight and obesity
* Hypertension
* Previous use of levothyroxine, antiepileptic drugs, or cardiac drugs within the last 6 months.
* Arrhythmia.
* Congenital or acquired heart disease
* Liver or kidney disease
* Hyperlipidemia
* Diabetes
* Infectious diseases
* Respiratory diseases
* Malignancies

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-05-24 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of left ventricle systolic function | 3 months post-procedure
  Left ventricle systolic function will be measured using left ventricle (LV) ejection fraction (LV EF%) where: (LV EF%) = (LVEDD)³ - (LVESD) / (LVEDD)³×100% LVEDD=left ventricular end-diastolic dimension. LVESD=left ventricular end-systolic dimension. LVFS=LV fractional shortening.

SECONDARY OUTCOMES:
Assessment of left ventricle fractional shortening | 3 months post-procedure
  Left ventricle fractional shortening (LV FS) will be measured. where: LV FS= LVEDD-LVESD/LVEDD X 100%.
  LVEDD=left ventricular end-diastolic dimension. LVESD=left ventricular end-systolic dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.